CLINICAL TRIAL: NCT03427281
Title: Postoperative Bracing Patterns After Lumbar Surgery for Degenerative Conditions in Belgium
Brief Title: Postoperative Bracing Patterns After Lumbar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KU/UZ Leuven S60109
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2020-02

CONDITIONS: Lumbar Spine Degeneration; Arthrosis; Spine; Surgery
MeSH Terms: conditions — Osteoarthritis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Masking Description: the investigator is blinded for the identity of the participating surgeons in the questionnaire
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort: Belgian orthopaedic surgeons & neurosurgeon (Experimental)
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — questionnaire to assess the patterns of postoperative bracing use by spinal surgeons in Belgium

SUMMARY:
A variety of postoperative bracing are routinely applied after spinal procedures but there are limited data regarding their efficacy, especially with the increasing use of internal fixation.Currently, no data are available regarding the use of postoperative braces in Belgium. Bracing is sometimes considered after lumbar surgery for degenerative conditions. All neurosurgeons and orthopedical surgeons in Belgium will be questioned to assess the patterns of postoperative bracing use after lumbar surgery.

DETAILED DESCRIPTION:
Subjects: all neurosurgeons and orthopedical surgeons in Belgium

Outcomes: The content of the questionnaire is based on a previously conducted study in the USA, cfr. "Bible, J. E., Biswas, D., Whang, P. G., Simpson, A. K., Rechtine, G. R., Grauer, J. N. (2009). Postoperative bracing after spine surgery for degenerative conditions: a questionnaire study. The Spine Journal, 9(4), p. 309-316." Permission to use this questionnaire was received from the corresponding author.

More specifically, a single-page questionnaire will be distributed to all spinal surgeons affiliated to the Spine Society Belgium. The questionnaire will focus on whether surgeons typically immobilize patients after specific spinal procedures, the type of orthosis used, the duration of treatment, and the rationale for bracing.

Data analysis: Both descriptive and inferential statistical methods will be used. The study Frequencies and percentages for categorical variables will be calculated. Chi-square analysis will be used. Significance level will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic surgeon or neurosurgeon in Belgium

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Whether or not surgeons typically immobilize patients after specific spinal surgical procedures | 2 months
  yes/no
Duration to prescribe a spinal orthosis after specific spinal surgical procedures | 2 months
  < 3 weeks, 3-8 weeks, 2-4 months, or > 4 months
Rationale to prescribe a spinal orthosis after specific spinal surgical procedures | 2 months
  to increase fusion rate, to improve pain, and/or to slow down the patient
Type of spinal orthosis prescribed after specific spinal surgical procedures | 2 months
  lumbar corset, off the shelf lumbosacral orthosis, and/or costum molded lumbosacral orthosis

CONTACTS AND LOCATIONS:
Overall Officials: Bart Depreitere, PhD, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Thijs Swinnen, MSc, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Tinne Thys, MSc, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Wim Dankaerts, PhD, PT, Principal Investigator — KU Leuven; Simon Brumagne, PhD, PT, Principal Investigator — KU Leuven; Peter Van Wambeke, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Lieven Moke, PhD, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Sebastiaan Schelfaut, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Ann Spriet, PT, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Lotte Janssens, PhD, PT, Principal Investigator — Hasselt University
Locations (1):
- UZ/KU Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bible JE, Biswas D, Whang PG, Simpson AK, Rechtine GR, Grauer JN. Postoperative bracing after spine surgery for degenerative conditions: a questionnaire study. Spine J. 2009 Apr;9(4):309-16. doi: 10.1016/j.spinee.2008.06.453. Epub 2008 Sep 14. PMID 18790685
- [Result] Bogaert L, Van Wambeke P, Thys T, Swinnen TW, Dankaerts W, Brumagne S, Moke L, Peers K, Depreitere B, Janssens L. Postoperative bracing after lumbar surgery: a survey amongst spinal surgeons in Belgium. Eur Spine J. 2019 Feb;28(2):442-449. doi: 10.1007/s00586-018-5837-0. Epub 2018 Nov 28. PMID 30488116